CLINICAL TRIAL: NCT06488885
Title: The Effect of Elderly Care Training Given to Nursing Students on Ageism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Ülkü YILMAZ, PHD, University of Beykent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2024/27
Record Dates: First submitted 2024-05-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Ageism
Keywords: "Nursing"; "Elderly Care"; "Ageism"
MeSH Terms: conditions — Ageism

STUDY DESIGN:
Intervention Model Description: This research was conducted at a foundation university's nursing school. The elderly care training given to students regarding ageism a randomized controlled study was conducted to determine the effect of It was designed as.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): Nursin students
  Interventions: Behavioral: Elderly care training
- Control group (No Intervention): Nursin students

INTERVENTIONS:
Behavioral: Elderly care training — The 60 experimental group students included in the study will have three lesson hours each week. Face-to-face training will be provided. Their consent was obtained before training was given to the experimental group. Participant Information Form and Positive and Negative Ageism Scale (PNYAÖ) will be applied as a pre-test. Trainings are 3 lesson hours, one day a week. It will be given as eight weeks and 24 hours in total. Upbeat and positive after the end of the training A posttest will be administered with the Negative Ageism Scale (PNSAS). Posttest PNSAÖ will be administered again one month after administration, and follow-up data will be obtained. Participant Information Form and Positive and Negative Ageism Scale (PNSAS) will be applied as a pre-test. Eight weeks. At the end, PNCAS will be administered again as the final test.
  Arms: Experimental group

SUMMARY:
geism is a multidimensional term that includes different attitudes, prejudices, behaviors and actions shown to a person simply because of his or her age. Today, in most societies in the world, elderly individuals are discriminated against. This discrimination stems from the negative attitudes of family members and society in general towards older individuals and aging. In most societies, old age and the changes that occur with aging are generally viewed negatively. Old age is seen as a process of decline in productivity, competence, individuality and independence in all areas of life. The elderly and old age can be viewed with stereotypes, prejudice and discrimination. Age discrimination includes beliefs and attitudes that can turn into discriminatory actions. Words synonymous with being old/aging generally carry negative content. These are generally negative situations such as dementia, weakness, disease, aging, deterioration, wear and tear, and inability to function. This research was designed as a randomized controlled study to determine the effect of elderly care training given to nursing students of a foundation university on their attitudes towards ageism. The population of the research consists of 150 first and second year nursing students of a foundation university in Istanbul between the 2023-2024 academic years. Power analysis was performed using the G*Power (v3.1.9) program to determine the sample size. It was calculated that there should be at least 26 participants in each group. The sample was planned with 120 students (60 experimental and 60 control groups) who met the study criteria and agreed to participate in the study. Number, percentage, mean and standard deviation will be used as descriptive statistical methods in the evaluation of the data. A normal distribution test will be applied to determine whether the research variables have a normal distribution. In case the research variables do not show normal distribution (p<0.05). In the analysis of variables for which the normality assumption is not met, non-parametric analysis methods Mann Whitney U (for comparisons of two groups) and Kruskal Wallis (for comparisons of three or more groups) will be used. Spearman correlation analysis will be performed to determine the relationship between the continuous variables of the research.

DETAILED DESCRIPTION:
The elderly population is increasing in our country. Türkiye Statistics According to the institution's data, the population aged 65 and over in our country in 2015 was 8.2% in 2023; this rate will increase to 10.2% in 2023 and 20% in 2050. It is predicted to increase to 20.8% and 27.7% in 2075. With the rapid increase in the elderly population, long life loneliness, poverty, disability, chronic diseases, care and support requirements, deterioration of health, and increase in addiction caused problems in maintenance. Psychophysiological problems and economic problems in elderly individuals The existence of difficulties has brought the issue of old-age services to the agenda. One of the difficulties experienced by the elderly is discrimination. Ageism is discrimination against a person simply because of their age. in the different attitudes, prejudices, behaviors, and actions shown. It is a multidimensional term that includes. Today In most societies around the world, elderly individuals are discriminated against is undergoing. This discrimination affects family members and society in general. As a result, their adverse effects on older individuals and aging stem from attitudes. In most societies, old age and Changes that occur with aging are generally negative is met. Aging is a decline in productivity, competence, individuality, and independence in all areas of life. İs observed. Stereotypes about old and old-age thoughts can be viewed with prejudice and discrimination. Old discrimination, beliefs, and attitudes can turn into discriminatory actions. It covers. Words synonymous with being old/aging generally contain harmful content. These are usually dementia, weakening, diseased, worn out, deteriorating, worn out, These are negative situations, such as the inability to function. In all societies, attitudes towards old age are generally positive and negative. Although they are mixed, the tendency for negative attitudes is greater. Society's and professionals' perceptions, perspectives, and perceptions of old age prejudices affect the quality of services provided to the elderly. Perception of old age; health Service in determining priorities in providing preventive health services in effectively implementing healthcare services for the elderly. Transportation, healthcare professionals in the field of elderly health In their specialization, policies towards old age can be effectively implemented directly or indirectly, impacting the problems experienced in its implementation. Negative attitudes towards elderly individuals in family life and society

There are some things that nurses should do to eliminate these attitudes:

There are applications. One of these applications is to help family members, and society understand that old age is a natural process that occurs during this period. Providing training on possible changes. This is what was done. Changes in individuals' aging process result from training.

Better understanding and more positive attitudes towards elderly individuals. It is thought that it may have. Health personnel are different types of people, such as geriatrics staff working in the field and university students. Age discrimination was studied in sample groups. In the works Researching individuals living in society Recommended. Having positive and negative attitudes towards the elderly in terms of the elderly's self-perception in society and quality of life is essential.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research,
* Being over 18 years old,
* Being a nursing student,
* Not having received any training, course or course regarding elderly care

Exclusion Criteria:

* Being under 18 years old
* Each participant will be required to fill out the survey form once.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Positive and negative ageism scale | The scale will be administered to the participants "as a pre-test" before training is given. The training duration is 8 weeks. It will be administered as a "final test" one week after the training is given. The scales will be applied to both experimental
  University students, it consists of two subscales developed to measure attitudes towards ageism. It is a measuring tool. Positive Age Discrimination Sub-dimension, which is one of the sub-dimensions The dimension affects the positive discriminatory attitudes of university students towards older people. It measures. There are 13 items in this subscale of the scale. Scale The highest score that can be obtained from this sub-dimension in the application is 65, and the lowest score is 65. The higher the score to be obtained, the more positive the attitude towards older people. Indicates that the level is high. Another sub-dimension, the Negative Age Discrimination Sub-Dimension, measures students' negative discriminatory attitudes towards older people.
Participant information form | The scale will be administered to the participants "as a pre-test" before training is given. The training duration is 8 weeks. It will be administered as a "final test" one week after the training is given. The scales will be applied to both experimental
  Participant information form prepared by the researchers. A total of 10 questions about the socio-demographic characteristics of the students and elderly individuals.
  Contains.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Beyketn University, Beylikduzu, Cumhuriyet Mahallesi, Turkey (Türkiye)